CLINICAL TRIAL: NCT05379322
Title: The Use of Synovial Biopsies in Predicting Response to Biologic Therapy in Rheumatoid Arthritis Patients
Acronym: SYBRA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision of the local healthcare authority
Sponsor: Abu Dhabi Stem Cells Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT.006.1.1.SYBRA
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Synovial biopsy; Biologic therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Etanercept; Certolizumab Pegol; golimumab; Janus Kinase Inhibitors; tofacitinib; baricitinib; upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Anti-TNF) (Experimental): Rheumatoid arthritis patients that have failed DMARD therapy will undergo a synovial biopsy under ultrasound guidance and sterile technique. Upon analysis of the sample, patients that are falling into the diffuse myeloid phenotype will be assigned to receive anti-TNF medication at the discretion of the treating physician.
  Interventions: Drug: Anti-TNF
- Group B (JAK inhibitor) (Experimental): Rheumatoid arthritis patients that have failed DMARD therapy will undergo a synovial biopsy under ultrasound guidance and sterile technique. Upon analysis of the sample, patients that are falling into the lymphoid- myeloid phenotype will be assigned to receive JAK inhibitor medication at the discretion of the treating physician.
  Interventions: Drug: JAK inhibitor
- Group C (Anti-TNF or JAK inhibitor) (Experimental): Rheumatoid arthritis patients that have failed DMARD therapy will undergo a synovial biopsy under ultrasound guidance and sterile technique. Upon analysis of the sample, patients that are falling into the pauci-cellular phenotype will be randomized to either anti-TNF or JAK inhibitor medication 1:1.
  Interventions: Drug: Anti-TNF; Drug: JAK inhibitor

INTERVENTIONS:
Drug: Anti-TNF — Upon analysis of the sample, patients that are falling into specific phenotypes (diffuse myeloid or pauci-cellular phenotypes) will be assigned to receive anti-TNF as biologic DMARD medications.
  Other Names: Adalimumab, etanercept, certolizumab, or golimumab
  Arms: Group A (Anti-TNF); Group C (Anti-TNF or JAK inhibitor)
Drug: JAK inhibitor — Upon analysis of the sample, patients that are falling into specific phenotypes (lymphoid- myeloid or pauci-cellular phenotypes) will be assigned to receive JAK inhibitors as biologic DMARD medications.
  Other Names: Tofacitinib, baricitinib, or upadacitinib
  Arms: Group B (JAK inhibitor); Group C (Anti-TNF or JAK inhibitor)

SUMMARY:
SYBRA is an open-label, phase 3, randomized controlled clinical trial that aims to assess the use of synovial biopsies in predicting response to biologic therapy in patients with rheumatoid arthritis that have failed disease-modifying drugs. The project has the potential to help change the current practice by offering the best treatment option. The decision to choose the best treatment for a particular patient is especially important in the context of the growing number of therapies available as a first-line option and the lack of specific biomarkers to predict response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject should be capable of consent
* Age 18 and older
* Classified as rheumatoid arthritis as per EULAR/ACR criteria 2010
* Failed one DMARD (Methotrexate, leflunomide, Sulfalsalazine, hydroxychloroquine)
* Can be on steroid dose <7.5mg
* Quantiferon negative
* Hepatitis B, C negative
* No recent history (<5y) of malignancy

Exclusion Criteria:

* Overlap syndrome
* Previously treated with a biological medication
* Heart failure NYHA III/IV
* Active tuberculosis
* Active infections
* Previous history of DVT, PE, or Stroke
* Other significant comorbidities that will prevent them from taking any biologic medication as per EULAR guidelines on treating rheumatoid arthritis 2020.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in DAS28 score | Baseline, Visit 3 (12 weeks)
  Change in DAS28 score indicating remission compared to baseline in at least 50% of patients, where DS28<2.6 indicated remission.
  * DAS score: disease activity score, where <2.6 indicates remission, 2.6-3.2 low disease activity. 3.2-5.1 moderate disease activity; >5.1 high disease activity; higher values suggest worse outcomes.

SECONDARY OUTCOMES:
Change in HAQ score | Baseline, Visit 3 (12 weeks)
  Significant decrease in HAQ score compared to baseline.
  * HAQ (Health assessment questionnaire). Scores vary from 0-to 3. Higher scores are associated with worse outcomes.
Change in power Doppler activity | Baseline, Visit 3 (12 weeks)
  Change in power Doppler activity compared to a baseline where no power Doppler activity indicates remission. Measurement in Doppler activity on ultrasound using a grading system developed by EULAR.
  * Global EULAR-OMERACT Synovitis Score: scores range from 0-3 for each scanned joint. Higher scores correlate with worse outcomes.
Change in cellular phenotype | Baseline, Visit 3 (12 weeks)
  Change in cellular phenotype compared to baseline. Estimation of change in the number of inflammatory cells as per the grading criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gianina Statache, MD, Principal Investigator — Abu Dhabi Stem Cells Center; Rene A. Rivero Jimenez, PhD, Study Chair — Abu Dhabi Stem Cells Center
Locations (1):
- Abu Dhabi Stem Cells Center, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No